CLINICAL TRIAL: NCT05629507
Title: Effectiveness of Immersive Virtual Reality in Patients With Cancer Undergoing Chemotherapy: a Randomized Controlled Trial
Brief Title: Effectiveness of Immersive Virtual Reality in Patients With Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ASL Gallura - Ospedale Giovanni Paolo II (Other)
Responsible Party: Principal Investigator, Salvatore Ortu, Principal Investigator, ASL Gallura - Ospedale Giovanni Paolo II
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: VROM_01
Record Dates: First submitted 2022-10-04; First posted 2022-11-29 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Cancer; Chemotherapy Effect; Anxiety; Fatigue; Pain
Keywords: Virtual Reality; Cancer; Chemotherapy; Anxiety; Fatigue; Pain
MeSH Terms: conditions — Neoplasms; Anxiety Disorders; Fatigue; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Virtual Reality (Experimental): In the virtual reality arm, patients will use a Virtual Reality headset. The multimedia contents in VR, will have a video quality from 4K to 8K, 360 degrees, and High Definition audio stereo.
  Interventions: Device: Virtual Reality
- Narrative Medicine (No Intervention): In narrative medicine arm, patients will express their subjective experience regarding to the chemotherapy through writing. The experience will be written in free form by the patient and will cover both the cognitive, emotional and perceptual aspects. A nurse will always be available to guide the patient in the activity of expressing cognitive, emotional and perceptual contents.
- Standard Care (No Intervention): In control arm, patients will be free to choose different activities during the infusion of chemotherapy, such as conversation with nurses, doctors, trainees, reading, writing, watching television, listening to music or videos on their smartphone.

INTERVENTIONS:
Device: Virtual Reality — The Virtual Reality intervention will administer through the use of a Virtual Reality headset. The multimedia contents in VR, will have a video quality from 4K to 8K, 360 degrees, and HD audio stereo.
  The scenarios are classified into 12 categories: 1) Artistic cities (60 scenarios); 2) Africa (17 scenarios); 3) Hills (26 scenarios); 4) Rivers, lakes and waterfalls (43 scenarios); 5) Sardinia (13 scenarios); 6) Deserts (21 scenarios); 7) Beaches (20 scenarios); 8) Animals (20 scenarios); 9) Mountains (25 scenarios); 10) Concerts (21 scenarios); 11) Sea (24 scenarios); 12) submarine (20 scenarios).
  Arms: Virtual Reality

SUMMARY:
The goal of this clinical trial is to study the effects of Immersive Virtual Reality in patients with cancer undergoing chemotherapy.

The main questions it aims to answer are:

* Could the immersive virtual reality application prevents or reduces anxiety, prevents or reduces fatigue, prevents or reduces pain, improves therapeutic adherence, prevents or reduces adverse events, then cancer patients treated with narrative medicine, and then cancer patients in standard care only?
* Could the immersive virtual reality application show symptoms of cybersickness?

Participants will be randomly allocated with balanced allocation ratio 1: 1: 1 into three groups: 1) Virtual Reality group; 2) Narrative medicine group; 3) Standard care group.

In the virtual reality arm, patients will use a Virtual Reality headset. The multimedia contents in VR, will have a video quality from 4K to 8K, 360 degrees, and High Definition audio stereo.

In control arm, patients will be free to choose different activities during the infusion of chemotherapy, such as conversation with nurses, doctors, trainees, reading, writing, watching television, listening to music or videos on their smartphone.

In narrative medicine arm, patients will express their subjective experience regarding to the chemotherapy through writing. The experience will be written in free form by the patient and will cover both the cognitive, emotional and perceptual aspects. A nurse will always be available to guide the patient in the activity of expressing cognitive, emotional and perceptual contents.

Researchers will compare the Virtual Reality group, Narrative Medicine group, Standard care group, to see the effects regarding to anxiety, fatigue, pain, improves therapeutic adherence and adverse events.

DETAILED DESCRIPTION:
This study is a three-arms randomized controlled trial that will be conducted at St Giovanni Paolo II Hospital, Olbia (Italy), from July 2022 to November 2022. This RCT, is an open-label trial, longitudinal, pre-post test, with balanced allocation ratio 1: 1: 1, monocentric, in patients with cancer undergoing intravenous chemotherapy.

Patients will be randomly allocated into three groups: 1) Virtual Reality group; 2) Narrative Medicine group; 3) Standard Care group.

Primary outcome is Anxiety, measured with State-Trait Anxiety Inventory. Secondary outcomes are: 1) fatigue measured with Revised Piper Fatigue Scale; 2) pain measured with Visual Analogic Scale; 3) Adverse effects, measured as manifestation of nausea, vomiting, needle phobia; 4) Symptoms of cybersickness will be measured with Reality Symptom Questionnaire.The study will conduct in accordance with the ethical standards as laid down in the Declaration of Helsinki, with the protocol approved by the Ethics Committee (Trial registration number: RS 97/CE). A written informed consent will obtain from all patients included in the study.

In the virtual reality arm, patients will use a Virtual Reality headset. The multimedia contents in VR, will have a video quality from 4K to 8K, 360 degrees, and High Definition audio stereo.The Virtual Reality headset will administer through the use of a Virtual Reality headset.The multimedia contents in VR, will have a video quality from 4K to 8K, 360 degrees, and HD audio stereo.

The scenarios are classified into 12 categories: 1) Artistic cities (60 scenarios); 2) Africa (17 scenarios); 3) Hills (26 scenarios); 4) Rivers, lakes and waterfalls (43 scenarios); 5) Sardinia (13 scenarios); 6) Deserts (21 scenarios); 7) Beaches (20 scenarios); 8) Animals (20 scenarios); 9) Mountains (25 scenarios); 10) Concerts (21 scenarios); 11) Sea (24 scenarios); 12) submarine (20 scenarios).

In control arm, patients will be free to choose different activities during the infusion of chemotherapy, such as conversation with nurses, doctors, trainees, reading, writing, watching television, listening to music or videos on their smartphone.

In narrative medicine arm, patients will express their subjective experience regarding to the chemotherapy through writing. The experience will be written in free form by the patient and will cover both the cognitive, emotional and perceptual aspects. A nurse will always be available to guide the patient in the activity of expressing cognitive, emotional and perceptual contents.

ELIGIBILITY:
Inclusion Criteria:

* age> 18 years;
* diagnosis of cancer with indication for intravenous chemotherapy;
* cognitively able to participate;
* no significant acoustic deficit;
* no significant visual impairment;
* sufficient ability to write and read in Italian.

Exclusion Criteria:

* use of antipsychotic drugs;
* epilepsy;
* use of drugs or alcohol;
* metastatic cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-11-16 (Actual)

PRIMARY OUTCOMES:
Change is being assessed for Anxiety | Baseline, pre-intervention and immediately after the intervention
  Anxiety is assessed with State-Trait Anxiety Inventory.The minimum value is 20 and the maximum value is 80, whether higher scores mean a worsening of anxiety.

SECONDARY OUTCOMES:
Assessment of Fatigue | Baseline, pre-intervention and immediately after the intervention
  Fatigue is assessed with Revised Piper Fatigue Scale. The minimum value is 0 and the maximum value is 10, whether higher scores mean a worsening of fatigue.
Assessment of Pain | Baseline, pre-intervention and immediately after the intervention
  Pain is assessed with Visual Analogic Scale.The minimum total score is 0 and the maximum is 10, whether higher scores mean a worsening of pain.
Number of partecipants with Adverse effects | Baseline, pre-intervention and immediately after the intervention
  Adverse effects are assessed as number of partecipants with nausea, vomiting, needle phobia.
Number of partecipants with a therapeutic adherence | Baseline, pre-intervention and immediately after the intervention
  The therapeutic adherence is assessed as number of partecipants with a reduction,delay, or discontinuation of chemotherapy administration.

CONTACTS AND LOCATIONS:
Overall Officials: Salvatore Ortu, Dr, Principal Investigator — Oncology Unit, Giovanni Paolo II Hospital, Olbia,Italy
Locations (1):
- Salvatore Ortu, Olbia, Sassari, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Burrai F, Ortu S, Marinucci M, De Marinis MG, Piredda M. Effectiveness of Immersive Virtual Reality in People with Cancer Undergoing Antiblastic Therapy: A Randomized Controlled Trial. Semin Oncol Nurs. 2023 Aug;39(4):151470. doi: 10.1016/j.soncn.2023.151470. Epub 2023 Jul 16. PMID 37455151